CLINICAL TRIAL: NCT01754350
Title: Calorie-restricted, Ketogenic Diet and Transient Fasting vs. Standard Nutrition During Reirradiation for Patients With Recurrent Glioblastoma: the ERGO2 Study
Brief Title: Calorie-restricted, Ketogenic Diet and Transient Fasting During Reirradiation for Patients With Recurrent Glioblastoma
Acronym: ERGO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Tavarlin (Industry)
Responsible Party: Principal Investigator, Johannes Rieger, PD Dr. med., Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERGO2
Record Dates: First submitted 2012-12-14; First posted 2012-12-21 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Recurrent Glioblastoma
Keywords: ketogenic diet; glioma; fasting; reirradiation; nutrition
MeSH Terms: conditions — Glioblastoma; Glioma; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketogenic diet and transient fasting (Experimental): Calorie-restricted, ketogenic diet and transient fasting during reirradiation
  Interventions: Dietary Supplement: calorie-restricted ketogenic diet and transient fasting
- standard nutrition (Active Comparator): nutrition according to recommendations of the German society for nutrition during reirradiation
  Interventions: Dietary Supplement: standard nutrition

INTERVENTIONS:
Dietary Supplement: calorie-restricted ketogenic diet and transient fasting — On day 1-3 and day 7-9, restriction of carbohydrates to < 60 g and of calories to 21-23 kcal/kg per day, on day 4-6 fasting. On day 1-3 and 7-9, restriction of carbohydrates can be supported by the use of drinks provided by "Tavarlin".
  Arms: ketogenic diet and transient fasting
Dietary Supplement: standard nutrition — nutrition as recommended by the german society for nutrition, 30 kcal/kg per day
  Arms: standard nutrition

SUMMARY:
Increased glucose metabolism is characteristic for solid tumors. Thereby, glucose is important for the generation of ATP, supply of anabolic substrates and defense against reactive oxygen species in tumor cells. In preclinical models, restricting glucose availability using a ketogenic diet, calorie-restriction or transient fasting inhibits tumor growth.

Therefore, the purpose of the study is to evaluate whether a calorie-restricted, ketogenic diet and transient fasting can enhance the efficacy of reirradiation in patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* recurrence of a histologically confirmed glioblastoma or gliosarcoma
* at least 6 months after first surgery
* at least 6 months after first radiotherapy
* interdisciplinary recommendation for reirradiation
* karnofsky performance status >= 60, ECOG <= 2
* creatinine <= 2,0 mg/dl, urea <= 100 mg/dl
* ALAT, ASAT <= 7x upper normal limit

Exclusion Criteria:

* bowel obstruction, subileus
* insulin-dependent diabetes
* decompensated heart failure (NYHA > 2)
* myocardial infarction within the last 6 months, symptomatic atrial fibrillation
* severe acute infection
* malnutrition, cachexia
* other medical conditions that might increase the risk of the dietary intervention
* pregnancy
* uncontrolled thyroid function
* pancreatic insufficiency
* dementia or other clinically relevant alterations of the mental status which could impair the ability of the patient to apply to the diet or understand the informed consent of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Dr. Senckenberg Institute of Neurooncology, Frankfurt
  - University of Tuebingen, Tübingen

REFERENCES:
- [Derived] Voss M, Wenger KJ, von Mettenheim N, Bojunga J, Vetter M, Diehl B, Franz K, Gerlach R, Ronellenfitsch MW, Harter PN, Hattingen E, Steinbach JP, Rodel C, Rieger J. Short-term fasting in glioma patients: analysis of diet diaries and metabolic parameters of the ERGO2 trial. Eur J Nutr. 2022 Feb;61(1):477-487. doi: 10.1007/s00394-021-02666-1. Epub 2021 Sep 6. PMID 34487222
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Voss M, Wagner M, von Mettenheim N, Harter PN, Wenger KJ, Franz K, Bojunga J, Vetter M, Gerlach R, Glatzel M, Paulsen F, Hattingen E, Baehr O, Ronellenfitsch MW, Fokas E, Imhoff D, Steinbach JP, Rodel C, Rieger J. ERGO2: A Prospective, Randomized Trial of Calorie-Restricted Ketogenic Diet and Fasting in Addition to Reirradiation for Malignant Glioma. Int J Radiat Oncol Biol Phys. 2020 Nov 15;108(4):987-995. doi: 10.1016/j.ijrobp.2020.06.021. Epub 2020 Jun 30. PMID 32619561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketogenic Diet and Transient Fasting | Standard Nutrition
Started | 25 | 25
Completed | 20 | 22
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketogenic Diet and Transient Fasting | Standard Nutrition | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 71] | 58 [26 to 75] | 57 [26 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 20 | 18 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression-free-survival
Description: Progression-free-survival rates 6 months after reirradiation based on response assessment in neuro-oncology criteria (RANO)
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Ketogenic Diet and Transient Fasting | Standard Nutrition
Number analyzed (Participants) | 20 | 22
percentage of participants | 20 | 16

2. Secondary Outcome: Feasibility Measured as Median Number of Days on Diet Per Patient and Average Calorie and Carbohydrate Intake Per Day During Day 1-9
Description: Feasibility of the calorie-restricted, ketogenic diet and the transient fasting measured as median number of days on diet per patient and average calorie and carbohydrate intake per day during day 1-9
Time Frame: day 1-12
Reporting Status: Not Posted

3. Secondary Outcome: Safety and Tolerability as Defined as Number of Patients With Adverse Events
Description: Safety and tolerability of the calorie-restricted, ketogenic diet and the transient fasting as defined as number of patients with adverse events
Time Frame: day 1-12
Reporting Status: Not Posted

4. Secondary Outcome: Progression-free-survival
Description: progression-free-survival rates 1 month and 3 month after reirradiation
Time Frame: 1 month, 3 months
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Description: overall survival after the reirradiation
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Frequency of Seizures
Description: frequency of seizures at day 1-12
Time Frame: day 1-12
Reporting Status: Not Posted

7. Secondary Outcome: Ketosis
Description: urine and blood ketosis and metabolic parameters (glucose, insulin, IGF-1) during day 1-12
Time Frame: day 1-12
Reporting Status: Not Posted

8. Secondary Outcome: Quality of Life as Measured by the EORTC Quality of Life Questionnaire
Description: Quality of life at day 1-12 as measured by the EORTC Quality of Life Questionnaire
Time Frame: day 1-12
Reporting Status: Not Posted

9. Secondary Outcome: Depression
Description: depression as measured by SCL-90 at day 1-12
Time Frame: day 1-12
Reporting Status: Not Posted

10. Secondary Outcome: Attention
Description: attention as measured by d2-testing at day 1-12
Time Frame: day 1-12
Reporting Status: Not Posted

11. Secondary Outcome: Response
Description: response assessment 1 month after reirradiation
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All, even non-serious adverse events, were monitored at start of treatment until end of intervention at day 12 to assess procedure-specific adverse events. After day 12, the prespecified secondary end point and adverse event "epileptic seizures"), and all serious adverse events were documented until the end of the study of individual patients (until primary end points was reached).
Description: Few minor adverse events are not listed seperately because some of these occured in the same patients.
Arm/Group | Ketogenic Diet and Transient Fasting | Standard Nutrition
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 4/20 | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketogenic Diet and Transient Fasting (N=20) | Standard Nutrition (N=22)
epileptic seizure (Nervous system disorders) | 1 (1) | 2 (2)
Others (Nervous system disorders) | 3 (3) | 3 (3) — headache, nausea or possible epileptic seizures with short lasting aphasia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT01754350/Prot_SAP_000.pdf